CLINICAL TRIAL: NCT00312442
Title: Study of Photodynamic Therapy With WST09 in Patients With Recurrent or Persistent Localized Carcinoma of the Prostate Following Radiation Therapy
Brief Title: Phase II/III Study of WST09 in Prostate Cancer After Radiation Therapy
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: STEBA decided to develop WST11 that is soluble in aqueous solutions. The property of WST 11 make it safer and better candidate for therapeutic applications.
Sponsor: STEBA France (Industry)
Responsible Party: STEBA FRANCE, STEBA FRANCE
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEC/WST0512 66N/WST 2.21
Record Dates: First submitted 2006-03-30; First posted 2006-04-10 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-05

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer after radiation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- WST 09 (Experimental): Treatment with WST09-mediated VTP
  Interventions: Drug: Treatment with WST09 Vascular Photodynamic therapy

INTERVENTIONS:
Drug: Treatment with WST09 Vascular Photodynamic therapy

SUMMARY:
The aim of this clinical trial is to evaluate the efficacy and safety of the WST09-mediated vascular-targeted photodynamic therapy (VTP) in patients with localized prostate cancer recurrent after external radiation therapy or temporary (High Dose Rate, or HDR) brachytherapy.

DETAILED DESCRIPTION:
This is a multicentre, open labelled, phase II/III, 6-month clinical trial with an additional follow-up at Month 12, aiming to determine the efficacy and tolerability of the WST09-mediated VTP treatment. This treatment consists of an I.V. infusion of WST09 (2 mg/kg), in combination with per-cutaneous interstitial illumination using laser light (wavelength at 763nm) delivered through optical fibres positioned through the perineum in the prostatic lobes.

Patients who are eligible to participate in the study must have a clinically diagnosed positive biopsy of the prostate (up to stage T2b-N0-M0) diagnosed after external radiotherapy or temporary brachytherapy (no seeds), and present with increasing PSA levels on three consecutive occasions (at least 3 months apart) post-radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

Histologically proven localized prostate cancer after receiving external radiation therapy;

Exclusion Criteria:

Patients unwilling or unable to give informed consent; Patients who received or are receiving chemotherapy; Patients previously treated with HIFU, cryotherapy, other salvage treatments, or with a trans-urethral resection of the prostate (TURP); Patients whose previous radiation therapy caused extensive cystitis and/or proctitis.

Patients suspected of Disseminated Intravascular Coagulation (DIC). Patients with prior history of coronary artery disease, angina pectoris, myocardial infarction, coronary angioplasty or coronary artery bypass graft, severe valvulopathy, cardiac failure, artrial fibrillation and / or sustained arrhythmia.

Patients whose cardiac status does not allow general anesthesia. Patients with history of thromboses or thrombo-embolisms. Patients with history of stroke or transient ischemic attack.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-05; Primary Completion 2008-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Prostate biopsy results at Month 6 after treatment. | 6 months

SECONDARY OUTCOMES:
Percentage of positive cores in the biopsies prior to and 6 months after the WST09-mediated VTP. | 6 months
PSA levels taken periodically for 1 year after the procedure | Month 1,3,6 and 1 year
Hypoperfusion according to MRI at Week 1 after the procedure. | 1 week and Month 6
Calculated PSA velocity before and after WST09-mediated VTP. | Month 1,3,6 and 1 year
Nadir of the PSA after the WST09-mediated VTP compared with the nadir of PSA after radiation therapy | Month 1,3,6 and 1 year
To assess the safety and tolerability of WST09-mediated VTP treatment in this patient population | Day1,Day 7, Month1,3,6,and 12
  The evaluation of safety will be based on reported adverse events, changes in vital signs and laboratory tests from the Treatment Visit until the study is completed.

CONTACTS AND LOCATIONS:
Overall Officials: John Trachtenberg, MD FRCS(C), Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada